CLINICAL TRIAL: NCT01866397
Title: Pharmacokinetics of Cidofovir During Continuous Venovenous Hemofiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna (Other)
Responsible Party: Principal Investigator, Florian Thalhammer, a.o.Univ.-Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CIDOFOVIR_CVVH
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Cytomegalovirus Retinitis; Acute Renal Failure
Keywords: cidofovir; cvvh; renal replacement therapy; HCMV; Pharmacokinetics of cidofovir during CVVH; continuous venovenous hemofiltration
MeSH Terms: conditions — Cytomegalovirus Retinitis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cidofovir pharmacokinetics (Experimental): Patient received cidofovir due to clinical necessity (therapy resistant HCMV retinitis) while being on continuous hemofiltration. Pre- and postfilter plasma samples were taken at multiple timepoints during 24 hours.
  Interventions: Other: Cidofovir pharmacokinetics

INTERVENTIONS:
Other: Cidofovir pharmacokinetics — Blood samples were drawn before and 15, 30, 60, 120, 240, 360, 720 and 1440 minutes after the start of the cidofovir infusion. Plasma and ultrafiltration samples were collected from the outlet of the ultrafiltrate compartment of the hemofilter.

SUMMARY:
Cidofovir is an acyclic nucleotide analog with broad-spectrum antiviral activity against herpesviruses. Its potency in inhibiting HCMV has been shown in conventional in vitro studies. It is approved for the systemic treatment of human cytomegalovirus (HCMV) retinitis in patients with AIDS and as a second line therapy for HCMV infections not responding to ganciclovir or foscarnet.

In intensive care patients continuous venovenous haemofiltration (CVVH) is a well-established extracorporal renal replacement therapy with a high clearance rate.

Pharmacokinetic studies of antifungal agents in critically ill patients treated with CVVH are rare. Elimination of any given drug by renal replacement therapy is determined by several major factors which are membrane specific, due to physico-chemical properties of the drug and characteristics of the renal replacement technique used.

Study objective The trial is conducted to investigate the pharmacokinetics of cidofovir during CVVH in critically ill patients. It is suspected that Hemofiltration will influence cidofovir plasma levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* Suspected of proven HCMV infection
* Suspected or proven resistancy of HCMV to the first line therapy (ganciclovir / foscarnet).
* Continuous venovenous hemodiafiltration (CVVHDF) due to acute or chronic renal failure.

Exclusion Criteria:

* Known history of hypersensitivity to cidofovir or probenecid.
* An expected survival of less than three days.
* Known alcohol dependency, epilepsy, pregnancy or liver failure.
* Infection with a ganciclovir or foscarnet susceptible HCMV strain

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2002-03; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
AreaUnderCurve (AUC) | 24 hours
  AUC (plasma concentration) of cidofovir during 24 hours of hemofiltration

SECONDARY OUTCOMES:
half-life (t1/2) of cidofovir during hemofiltration | 24 hours
maximum and minimum plasma concentration (Cmax, Cmin) of cidofovir during hemofiltration | 24 hours
total body clearance (Cltot) of cidofovir during hemofiltration | 24 hours
hemofiltration clearance (ClHF) of cidofovir during hemofiltration | 24 hours
sieving coefficient of cidofovir during hemofiltration | 24 hours
elimination fraction of cidofovir during hemofiltration | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Florian Thalhammer, Prof. MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria